CLINICAL TRIAL: NCT04373512
Title: Intravesical Lactobacillus to Reduce Urinary Symptoms After Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001124
Record Dates: First submitted 2019-11-01; First posted 2020-05-04 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Neurogenic Bladder
Keywords: Intermittent Catheter
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Design: Prospective, randomized pilot intervention clinical trial. Target Enrollment: 182 subjects total at least 1-year post-SCI. Setting: National sample (N=114 intervention only, no urine collection) and local Washington, DC metropolitan area (N=68 intervention + urine collection).
  Controls: This is a 2-arm dose-finding pilot clinical trial, as such there is no control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dosage Group (Experimental): For the LGG® instillation, participants will be instructed to mix the contents of 1 LGG capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG mixture into a 60cc syringe and instill via the intermittent catheter. Participants will receive 2 LGG capsules and will repeat this process the following day ("Low" dose). Subjects will remain in the study for up to 29 months, with participation ending after one completed intervention (2 doses) and post-intervention assessments are complete. If urinary symptoms do not occur warranting instillation during the ensuing 29 months, participants will be asked to return any remaining kits (including LGG®). Participants will be instructed to complete the USQNB-IDC weekly until study completion.
  Interventions: Drug: Culturelle 10 Billion CFU Capsule (2 doses)
- High Dosage Group (Experimental): For the LGG® instillation, participants will be instructed to mix the contents of 1 LGG capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG mixture into a 60cc syringe and instill via the intermittent catheter. Participants will receive 4 LGG capsules and will repeat this process the following day twice for a total of four doses ("High" dose). Subjects will remain in the study for up to 29 months, with participation ending after one completed intervention (4 doses) and post-intervention assessments are complete. If urinary symptoms do not occur warranting instillation during the ensuing 29 months, participants will be asked to return any remaining kits (including LGG®). Participants will be instructed to complete the USQNB-IDC weekly until study completion.
  Interventions: Drug: Culturelle 10 Billion CFU Capsule (4 doses)

INTERVENTIONS:
Drug: Culturelle 10 Billion CFU Capsule (2 doses) — For the LGG instillation, participants will be instructed to mix the contents of 1 LGG capsule into saline. After mixing, participants will draw up the liquid LGG mixture into a syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Participants will receive 2 LGG capsules and will repeat this process the following night ("Low" dose). Subjects will remain in the study for up to 29 months, with participation ending after one completed intervention (2 doses) and post-intervention assessments are complete. If urinary symptoms do not occur warranting instillation during the ensuing 29 months, participants will be asked to return any remaining capsules
  Other Names: Lactobacillus RhamnosusGG
  Arms: Low Dosage Group
Drug: Culturelle 10 Billion CFU Capsule (4 doses) — For the LGG instillation, participants will be instructed to mix the contents of 1 LGG capsule into saline. After mixing, participants will draw up the liquid LGG mixture into a syringe and instill via the intermittent catheter after the last catheterization prior to going to bed. Participants will receive 4 LGG capsules and will repeat this process twice daily for a total of four doses ("High" dose). Subjects will remain in the study for up to 29 months, with participation ending after one completed intervention (4 doses) and post-intervention assessments are complete. If urinary symptoms do not occur warranting instillation during the ensuing 29 months, participants will be asked to return any remaining capsules
  Other Names: Lactobacillus RhamnosusGG
  Arms: High Dosage Group

SUMMARY:
The objectives of the proposed research among this population are: 1) to define clinically meaningful change (i.e. differentiating states of health and illness) with respect to urinary symptoms, urine inflammation, cultivable bacteria, and the urine ecosystem; and 2) to determine the optimal intravesical Lactobacillus RhamnosusGG (LGG®) dose to be used to reduce urinary symptoms in a future clinical trial.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is the most common outpatient infection world-wide, and for people with spinal cord injury (SCI) and neurogenic bladder (NB), it is the most common infection, secondary condition, cause for emergency room visits, and infectious cause of hospitalization. Despite its prevalence, attempts to ameliorate UTI among people with SCI are stymied by long-standing diagnostic challenges which arise from evidence gaps around "gold standard" diagnostic tests (urinalysis and urine culture) that have lower sensitivity and specificity for UTI in this population. A high prevalence of chronic inflammation leading to persistence of white blood cells (WBC) in the urine confounds the utility of WBC count, pyuria, and leukocyte esterase as biomarkers for UTI; nitrites in urine indicate the presence of only specific (but not all) organisms, many of which are present to a greater extent in the urine of people with SCI; and people with SCI have a high prevalence of asymptomatic bacteriuria. These physiologic changes render the gold standard diagnostic tests less useful for identifying UTI in persons with SCI.

SPECIFIC AIM 1

2 urine samples (sampling at least 2 weeks apart) for urinalysis, urine culture, uNGAL, and NGS (16S rRNA and shotgun) under the same conditions. In addition to completing the USQNB-IC prior to urine collection, participants will complete the USQNB-IC 3 days after urine collection

SPECIFIC AIM 2 Intravesical LGG dose (group: high or low) will be obtained, USQNB-IC, urine collection for urinalysis, culture, NGAL and next generation sequencing as described above. And patient satisfaction questions.

ELIGIBILITY:
Inclusion Criteria:

* SCI at least 1-year duration;
* Neurogenic bladder;
* Utilizing intermittent catheterization for bladder management;
* Women must be premenopausal and not currently menstruating;
* Community dwelling

Exclusion Criteria:

* Use of prophylactic antibiotics;
* Instillation of intravesical antimicrobials to prevent UTI;
* Psychologic or psychiatric conditions influencing the ability to follow instructions;
* Use of oral or IV antibiotics within the past 2 weeks;
* Sexual activity within the previous 72 hours;
* Participation in another study with which results could be confounded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA1) day of urine collection
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA1) day 1 post urine collection
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA1) day 2 post urine collection
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA1) day 3 post urine collection
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA2) Weekly up to 29 months
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA2) day 1 of intervention
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Urinary Symptom Questionnaire for Neurogenic Bladder- Intermittent catheter | (SA2) 24-48 hours after intervention completion
  Will measure change in urinary symptoms for those that use an intermittent catheter. Higher scores may mean worse outcomes.
Change in Urine white blood cell count | (SA1) day 1 post urine collection
  urinalysis
Change in Urine white blood cell count | (SA1) day 14 post urine collection
  urinalysis
Change in Urine white blood cell count | (SA 2) day 1 of intervention
  urinalysis
Change in Urine white blood cell count | (SA 2) 24-48 hours after intervention completion
  urinalysis
Change in Urine Nitrite | (SA1)day 1 post urine collection
  urinalysis
Change in Urine Nitrite | (SA1)day 14 post urine collection
  urinalysis
Change in Urine Nitrite | (SA 2) day 1 of intervention
  urinalysis
Change in Urine Nitrite | (SA 2) 24-48 hours after intervention completion
  urinalysis
Change in Urine NGAL | (SA1)day 1 post urine collection
  Urine NGAL
Change in Urine NGAL | (SA1)day 14 post urine collection
  Urine NGAL
Change in Urine NGAL | (SA 2) day 1 of intervention
  Urine NGAL
Change in Urine NGAL | (SA 2) 24-48 hours after intervention completion
  Urine NGAL
Change in Cultivable Bacteria | (SA1)day 1 post urine collection
  urine culture
Change in Cultivable Bacteria | (SA1)day 14 post urine collection
  urine culture
Change in Cultivable Bacteria | (SA 2) day 1 of intervention
  urine culture
Change in Cultivable Bacteria | (SA 2) 24-48 hours after intervention completion
  urine culture
Change in Urine microbiome composition | (SA1)day 1 post urine collection
  proportion of different bacterial species
Change in Urine microbiome composition | (SA1)day 14 post urine collection
  proportion of different bacterial species
Change in Urine microbiome composition | (SA 2) day 1 of intervention
  proportion of different bacterial species
Change in Urine microbiome composition | (SA 2) 24-48 hours after intervention completion
  proportion of different bacterial species
International SCI Lower Urinary Tract Function Basic Data Set | Day 1
  A tool to describe urinary tract impairment, awareness of need to empty the bladder, main bladder emptying method, medications used for bladder management, surgeries, and change in urinary symptoms in the past year. Score is not associated with outcome
International SCI Core Data Set | Day 1
  Includes date of injury, dates of initial hospitalization admission and discharge, neurological data. Score is not associated with outcomes
NINDS Medical History CDE: | Day 1
  A brief medical history using body system categories. Score is not associated with outcomes
NINDS Prior and Concomitant Medications CDE | Day 1
  Contains whether or not the participant is taking a medication during the study protocol, name of medication, reason for medication, medication dose, frequency, start and end dates, and free text. Score is not associated with outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Groah, MD, MSPH, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No